CLINICAL TRIAL: NCT06709040
Title: A Non-interventional, Observational, Registry-based Study to Investigate Long-term Safety and Clinical Parameters of Somapacitan Treatment in Paediatric Patients With Growth Hormone Deficiency During Routine Clinical Practice
Brief Title: A Study to Follow Paediatric Participants With Growth Hormone Deficiency Treated With Somapacitan for Long Term Safety Information and Clinical Parameters
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8640-4787; U1111-1294-5941 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Growth Hormone Deficiency; Neoplasms; Diabetes Mellitus Type 2
MeSH Terms: conditions — Dwarfism, Pituitary; Neoplasms; Diabetes Mellitus, Type 2 | interventions — somapacitan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Growth Hormone Deficieny: The study is non-interventional as there are no interventions involved and decision to treat participants with commerically available somapacitan will be made at the treating physician's discretion prior to, and independently from, the decision to include the participants in the GLoBE-Reg registry. Novo Nordisk will not provide any products for included participants during the conduct of the study.
  Interventions: Drug: Somapacitan

INTERVENTIONS:
Drug: Somapacitan — Participants will be treated with commercially available somapacitan according to routine clinical practice at the discretion of the treating physician.

SUMMARY:
The aim of this study is to look at the long-term safety and clinical parameters of somapacitan in paediatric participants with growth hormone deficiency under routine clinical practice conditions. The study population will include 400 paediatric growth hormone deficient participants from the Global Registry for Novel Therapies in Rare Bone and Endocrine Conditions (GloBE-Reg) treated with once-weekly somapacitan and fulfilling the eligibility criteria of the study. The total duration of the study is planned to 10 years consisting of a 5-year recruitment period in the GLoBE-Reg followed by a 5-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Treated with commercially available somapacitan according to local practice at the discretion of the physician.
* Primary confirmed diagnosis of growth hormone deficiency as per local practice.
* Male or female below 18 years of age at the time of signing informed consent in the GLoBE-Reg.

Exclusion Criteria:

* Participants with active malignancy or in treatment for active pre-existing malignancy.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Paediatric participants with growth hormone deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2034-04-14 (Estimated); Study Completion 2034-04-14 (Estimated)

PRIMARY OUTCOMES:
Number of adverse drug reactions | From baseline (week 0) to end of study (up to 10 years)
  Measured as count of events.

SECONDARY OUTCOMES:
Number of medication errors (incorrect dose administration) | From baseline (week 0) to end of study (up to 10 years)
  Measured as count of errors.
Number of participants with incident neoplasm | From baseline (week 0) to end of study (up to 10 years)
  Measured as number of participants (yes/no).
Number of participants with incident diabetes mellitus type 2 | From baseline (week 0) to end of study (up to 10 years)
  Measured as number of participants (yes/no).
Height velocity | From baseline (week 0) to end of study (up to 10 years)
  measured as centimeter per year (cm/year).
Change in height velocity standard deviation score (HVSDS) | From baseline (week 0) to end of study (up to 10 years)
  Measured as score ranging from -10 to +10.
Change in height standard deviation score (HSDS) | From baseline (week 0) to end of study (up to 10 years)
  Measured as score ranging from -10 to +10.
Change in insulin-like growth factor I (IGF-I) standard deviation score (SDS) | From baseline (week 0) to end of study (up to 10 years)
  Measured as score ranging from -10 to +10.
Change in bone age (measured as years) | From baseline (week 0) to end of study (up to 10 years)
  Measured as years.
Change in bone age (measured as months) | From baseline (week 0) to end of study (up to 10 years)
  Measured as months.
Participants reaching near adult height | at 10 year
  Near adult height defined as: height velocity <2 cm/year over the last 9 months and chronological age >16 years (males) or >15 years (females) or bone age >16 years (males) and > 15 years (females). Measured as number of participants (yes/no). Only for those who are expected to reach near adult height during the study.
Change in height SDS in participants reaching near adult height | From baseline (week 0) to end of study (up to 10 years)
  Near adult height can be defined as: height velocity <2 cm/year over the last 9 months and chronological age >16 years (males) or >15 years (females) or bone age >16 years (males) and > 15 years (females). Measured as score ranging from -10 to +10. Only for those who are expected to reach near adult height during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- University of Glasgow, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisktrials.com